CLINICAL TRIAL: NCT00055952
Title: A Phase II Study Of Intravenous DX-8951f (EXATECAN MESYLATE) Administered Daily For Five Days Every Three Weeks To Pediatric And Young Adult Patients With Ewing's Sarcoma (ES), Primitive Neuroectodermal Tumor (PNET), Or Desmoplastic Small Round Cell Tumor (DSRCT)
Brief Title: Exatecan Mesylate in Treating Patients With Ewing's Sarcoma, Primitive Neuroectodermal Tumor, or Desmoplastic Small Round Cell Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271889; DAIICHI-8951A-PRT034; SJCRH-DXEWS
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Sarcoma
Keywords: childhood desmoplastic small round cell tumor; metastatic childhood soft tissue sarcoma; nonmetastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Desmoplastic Small Round Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of exatecan mesylate in treating patients who have relapsed or refractory Ewing's sarcoma or peripheral primitive neuroectodermal tumor or desmoplastic small round cell tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with Ewing's sarcoma, primitive neuroectodermal tumor, or desmoplastic small round cell tumor treated with exatecan mesylate.
* Determine the time to tumor progression in patients treated with this drug.
* Determine median survival and 6- and 12-month survival of patients treated with this drug.
* Determine the pain response in patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, non-randomized, multicenter study. Patients are stratified according to disease (relapsed or refractory localized or metastatic Ewing's sarcoma or primitive neuroectodermal tumor vs desmoplastic small round cell tumor).

Patients receive exatecan mesylate IV over 30 minutes on days 1-5. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity for a maximum of 12 courses, or 6 courses beyond maximal response (whichever is longer).

Patients are followed every 3 months for 1 year after withdrawal from study.

PROJECTED ACCRUAL: A total of 13-27 patients will be accrued for stratum I within 12 months. A total of 9-17 patients will be accrued for stratum II within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically confirmed diagnoses:

  * Relapsed or refractory Ewing's sarcoma or primitive neuroectodermal tumor
  * Desmoplastic small round cell tumor
* Measurable disease

  * The following are not considered measurable disease:

    * Ascites
    * Pleural effusion
    * Lytic bone lesions
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2 (over 10 years of age)
* Lansky 60-100% (10 years of age and under)

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 750/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 8.5 g/dL

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST or ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Albumin at least 2.8 g/dL

Renal

* Creatinine less than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active serious infection
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No overt psychosis or mental disability that would preclude informed consent
* No other life-threatening illness within the past 6 months

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior autologous bone marrow or stem cell transplantation
* No concurrent biologic therapy

Chemotherapy

* Recovered from prior systemic chemotherapy
* Prior topoisomerase I inhibitor therapy allowed
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior cranial, spinal, or whole pelvis radiotherapy
* More than 4 weeks since prior radiotherapy to 25% of bone marrow reserve
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior major surgery and recovered
* No concurrent surgery

Other

* More than 28 days since prior investigational drugs (including analgesics or antiemetics)
* No more than 2 prior treatment regimens for this disease
* No other investigational drugs during and for 28 days after study therapy
* No other concurrent anticancer therapy
* No concurrent grapefruit or grapefruit juice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (9):
- United States (8):
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada